CLINICAL TRIAL: NCT04320966
Title: Neurovascular Complications and White Matter Damage in Acquired Anemias
Status: Withdrawn | Type: Observational
Why Stopped: Study was not funded.
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, John C. Wood, Professor, Children's Hospital Los Angeles
Other Study IDs: CHLA-20-00037
Record Dates: First submitted 2020-03-16; First posted 2020-03-25 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Anemia; Iron-deficiency Anemia; Healthy Controls
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Acquired Anemia: Otherwise healthy individuals with hemoglobin below 10.5 g/dl or hematocrit below 32
- Control: Age and sex matched individuals with hemoglobin in the upper quartile of normal

SUMMARY:
This is an observational trial, in patients with moderate to severe anemia and control subjects. The main purpose of this study is to understand whether normal brain blood flow, oxygen extraction reserve, white matter volumes, and brain functional connectivity are affected by acquired anemia. The investigators will perform baseline MRI monitoring for all subjects. All eligible subjects will be asked to provide informed consent before participating in the study.

DETAILED DESCRIPTION:
This is an observational trial, in patients with moderate to severe anemia and control subjects. The main purpose of this study is to understand whether normal brain blood flow, oxygen extraction reserve, white matter volumes, and brain functional connectivity are affected by acquired anemia. The investigators will perform baseline MRI monitoring for all subjects. All eligible subjects will be asked to provide informed consent before participating in the study. Comprehensive cerebrovascular MRI, baseline bloodwork, and neurocognitive testing will be collected from all subjects.

ELIGIBILITY:
Inclusion criteria (observational component):

* Age between 16 and 60 years of age.
* Any ethnicity.
* Either sex.
* Anemic group: hemoglobin less than 10.5 g/dl on screening hemoglobin.
* Control group: hemoglobin >13.2 g/dl for females, >14.6 g/dl for males, comparable age, sex and ethnicity to currently enrolled anemic subjects.

Exclusion criteria (observational component):

* Diabetes requiring medication.
* Hypertension requiring medication.
* Sleep disordered breathing requiring intervention.
* Body mass index >35 (morbid obesity)
* Contraindications to MRI, including pacemaker, severe claustrophobia, pregnancy.
* Known systemic inflammatory disease such as inflammatory bowel disease, systemic lupus erythematosus, or scleroderma.
* Known HIV.

Inclusion criteria (interventional component):

* Criteria for observational component, plus
* ron deficiency anemia based upon attending hematologist interpretation of transferrin saturation, ferritin, and other ancillary labs including hs-CRP, MMA.

Exclusion criteria (interventional component):

* Criteria for observational component, plus
* Prior reaction to intravenous iron.
* History of multiple drug allergies.
* History of severe asthma, eczema, or atopy.
* Systemic mastocytosis.
* Severe respiratory or cardiac disease.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Anemic subjects from Blood Donor Centers across Los Angeles will be recruited, the abnormal Menstrual Bleeding Clinic at Children's Hospital Los Angeles, and from the community if anemia can be documented.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Impact of acquired anemia on cerebrovascular oxygen delivery (ml O2/100g/min) | Day 0
  Impact of acquired anemia on cerebrovascular oxygen delivery will be assessed by measuring cerebral blood flow and oxygen content through MRI.
Impact of acquired anemia on cerebrovascular flow reactivity (%SI change/%ETCO2) | Day 0
  baseline MRI with blood oxygenation level dependent (BOLD) acquisition will be assessed in response to carbon dioxide exposure to determine whether acquired anemia affects cerebrovascular reserve
Impact of acquired anemia on blood brain barrier permeability surface area product (ml H20/100g/min) | Day 0
  baseline PSA product using water-extraction-with-phase-contrast-arterial-spin-tagging (WEPCAST) MRI will be assessed to determine whether acquired anemia affects blood brain barrier permeability to water
Impact of acquired anemia on cerebral metabolic rate of oxygen (ml O2/100g/min) | Day 0
  T2 relaxation under spin tagging (TRUST) acquisition via MRI will be used to assess any impact of anemia on cerebral metabolic rate of oxygen.
Impact of acquired anemia on total brain blood flow (ml blood/100g/min) | Day 0
  Phase contrast MRI will be assessed to determine whether acquired anemia affects total brain blood flow

CONTACTS AND LOCATIONS:
Overall Officials: John Wood, MD,PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (4):
- United States (4):
  - City of Hope Blood Donor Center, Duarte, California
  - Cedar Sinai Blood Bank, Los Angeles, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California, Los Angeles Blood Donor Center, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No